CLINICAL TRIAL: NCT01793467
Title: Solid Organ Transplantation and the Use of Raltegravir in HIV-Infected Patients: An Observational Study of Pharmacokinetics, Safety, Tolerability and Efficacy
Brief Title: Transplantation and the Use of Raltegravir in HIV-Infected Patients
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00036598
Record Dates: First submitted 2013-02-13; First posted 2013-02-15 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-07

CONDITIONS: HIV Positive; Organ Transplant Recipient; Active Wait Listing for Organ Transplant
MeSH Terms: conditions — HIV Seropositivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Raltegravir (RAL) is a preferred option for initial antiretroviral therapy in the most recent HIV Treatment Guidelines and is emerging as a popular choice for use in the specialized population of HIV-infected patients being considered for solid organ transplantation. Data from HIV-infected persons with normal organ function have revealed few raltegravir-associated metabolic complications compared to older antiretrovirals, and in general, drug-drug interactions with raltegravir are infrequent. The absence of such concerns appears to make raltegravir a potentially appealing option for antiretroviral therapy in HIV-infected patients being considered for solid organ transplantation.

At present, however, little is known of the safety and long term tolerability of RAL-containing regimens in persons undergoing solid organ transplantation. As more HIV-infected patients undergo organ transplantation, there is a growing need for good data on such things as the effect of dialysis on RAL concentrations, the potential interactions with commonly used immunosuppressive drugs, and the pharmacokinetic (PK) /pharmacodynamic (PD) characteristics in those with end stage organ failure, as well as those with functioning grafts.

The proposed study will also examine transplant function and survival in HIV-infected patients receiving RAL-containing ART and will compare it to HIV negative historic controls.

DETAILED DESCRIPTION:
Pre-transplant:

* Patients on stable antiretroviral regimens who undergo evaluation for transplantation and are subsequently placed on the transplant waiting list will be considered for inclusion in the study. The details of the cART for each patient will remain the sole purview of the patient and the patient's HIV care provider.
* To be considered for solid organ transplantation, in addition to routine transplant listing criteria, the patient must fulfill the following criteria:

  1. non-pregnant adult patient with CD4 count >200/μL;
  2. no concurrent active AIDS-defining infections or malignancy;
  3. at least 24 months of well controlled HIV viremia, defined as <50 copies for the majority of the time.

After all screening procedures have been completed to ensure eligibility, a pre-transplant pharmacokinetic study will be done as described below. Using specimens obtained during 7 time points, patient-specific Cmax, Cmin and AUC determinations will be made using standard calculation approaches. The PK data will also include samples drawn on dialysis days for patients with End-stage renal failure:- pre-dialysis, arterial and venous concentrations (Cin and Cout) at the beginning of dialysis, and post dialysis levels (to determine individual hemodialysis extraction ratios).

Additional data to be collected include a Quality of Life questionnaire, SF-36, and a PHQ-9 depression screen which will be administered as a baseline test done at enrollment. Patients will be asked to have a dual-emission X-ray absorptiometry (DEXA) scan prior to transplant (unless this has been completed within two years of enrollment).

Peri-transplant Assessments:

In addition to the standard of care laboratory and imaging procedures that are done around the time of organ transplantation, the following research samples will be collected:

* Pre-transplant - RAL concentrations
* In addition, the following information will be recorded from the subject's medical record: full HIV and infective history and test results including CD4 count, and percentage, HIV viral load, electrocardiography (to assess QTc interval), CMV-IgG/IgM, Hepatitis B, C, D screens +/- viral loads if not already determined.

Post-transplant inpatient hospitalization

* RAL concentrations as well as HIV viral load and CD4/CD8 lymphocyte populations.
* In addition, the following information will be recorded from the subject's medical record: test results including EKG (to assess QTc interval).

Post-transplant:

* RAL concentrations will be collected at Months 1 and 3 only.
* In addition to the routine post-transplant care, the following information will be collected from the subject's medical records at study months 1, 3, 6, 9, 12, 24 post transplant: CD4 count and %, HIV viral load (+/- genotype and integrase mutation analysis if viral rebound occurs), Vitamin D, Basic Metabolic Panel (to calculate ClCr), quantitative urinary creatinine and protein excretion. Patient side-effect card will be ascertained by directed questioning from the study coordinator at each visit.

Repeat DEXA scan will be done at the 24 months post-transplant visit. Quality of Life assessment and depression screening tools will be administered at the 6 and 24 month marks.

ELIGIBILITY:
Inclusion Criteria:

1. non-pregnant adult patient with CD4 count >200/μL
2. no concurrent active AIDS-defining infections or malignancy
3. at least 24 months of well controlled HIV viremia, defined as <50 copies for the majority of the time.
4. otherwise suitable transplant candidates, actively listed
5. currently taking Raltegravir for control of HIV infection

Ages: 13 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HIV positive patients, awaiting or listed for organ transplantation, currently taking Raltegravir
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
To examine raltegravir (RAL) in the management of HIV-infected persons listed for solid organ transplantation, with a focus on mortality and graft survival | 3+ years

SECONDARY OUTCOMES:
Assess Raltegravir viability as a long term HIV treatment drug for patients undergoing transplant | 3+ years
  1. Characterize the effect of raltegravir-based regimens on the pre and post-transplant endocrine and cardiovascular effects
  2. Evaluate drug-drug interactions between raltegravir and current transplant immunosuppressant regimens.
  3. Determine RAL pharmacokinetic (PK) profile in HIV-infected patients with end organ failure before and after organ transplantation.
  a) Measure RAL PK in HIV-infected patients with end-stage renal failure (ESRF), who are receiving dialysis pre-transplant.
  b) Assess raltegravir PK in patients with different severities of liver disease, including cirrhosis, when such patients are available.
  d) Assess the ability of RAL-centered ART combinations to maintain HIV suppression and CD4 counts following solid-organ transplant.
determine the viability of grafted organs in patients with HIV infections | 3+ years
  1. Track adverse events including those attributable to ART therapy, but also routine post-transplant events. Assess the safety and tolerability profile of RAL during the pre and post-transplant period.
  2. Determine graft survival and performance following transplantation in this population and compare to similar data in HIV-negative historical controls.

CONTACTS AND LOCATIONS:
Overall Officials: Cameron R Wolfe, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States